CLINICAL TRIAL: NCT07045948
Title: Biannual Review of Exhaled Air and Trends in Health Evaluation in COPD
Acronym: BREATHE-COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25213_BREATHE-COPD
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-06

CONDITIONS: COPD
Keywords: FeNO; Blood eosinophil count; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm: Stable COPD Patients with Longitudinal FeNO and Blood Eosinophil Monitoring (Other)
  Interventions: Diagnostic Test: Blood eosinophil Count

INTERVENTIONS:
Diagnostic Test: Blood eosinophil Count — Blood sample for blood eosinophil count

SUMMARY:
This study aims to evaluate how airway inflammation, lung function, and symptoms change over time in people with chronic obstructive pulmonary disease (COPD). Airway inflammation will be assessed using a simple breath test (FeNO) and a small blood sample to measure eosinophils, a type of white blood cell. Participants will be followed for one year, with three study visits (at the start, 6 months, and 12 months). The goal is to understand how these markers evolve and whether they differ between people who experience a worsening of symptoms (called exacerbations) and those who remain stable. All tests except for a small extra blood draw are part of routine COPD care. Participation does not affect standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 40 years
* Diagnosed with COPD according to GOLD criteria
* Attending routine follow-up visits every 6 months
* Ability to provide informed consent

Exclusion Criteria:

* Recent respiratory tract infection or exacerbation (either moderate or se-vere) (<4 weeks before inclusion)
* Dominant asthmatic phenotype (ACO with asthma predominance)
* Severe comorbidities interfering with participation or follow-up

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the longitudinal stability of FeNO levels in COPD patients over a 12-month period with biannual measurements. | from enrollment to the end of the study period (1 year)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: Undecided